CLINICAL TRIAL: NCT06630923
Title: HUMAN ALBUMIN IN HEART FAILURE - DIORASIS TRIAL
Brief Title: PREVENTION OF WORSENING RENAL FUNCTION OF INTRAVENUS ALBUMIN IN HEART FAILURE PATIENTS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Marios-Vasileios Koutroulos, Cardiology Resident, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6/ 29.2.2016
Record Dates: First submitted 2023-03-29; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Diuretics Drug Reactions; Heart Failure; With Decompensation; Albumin; Double
Keywords: Human Albumin; Furosemide; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Human Albumin + IV Furosemide (Active Comparator): Continuous slow IV infusion of Human Albumin plus IV Furosemide
  Interventions: Drug: Human albumin
- IV Furosemide alone (Placebo Comparator): Continuous slow IV infusion of Furosemide
  Interventions: Drug: Human albumin

INTERVENTIONS:
Drug: Human albumin — Experimental intervention (Group A): Continuous slow IV infusion of Human Albumin, based on diuresis-adjusted dosing, not later than 30 minutes after randomisation and not later than 2 hours after admission. Concomitant continuous slow IV infusion of diuretics (furosemide) based on body weight- and diuresis-adjusted dosing. Control intervention (Group B): Continuous slow IV infusion of diuretics (furosemide), based on body weight - and diuresis-adjusted dosing. Experimental intervention (Human Albumin) is off-label treatment for patients with acute decompensation of CHF in Greece. Control intervention (IV diuretic therapy) is on-label treatment for acute decompensation CHF in Greece.

SUMMARY:
Patients hospitalized for acute decompensation of CHF are usually complicated by worsening renal function (WRF) which leads to diuretic resistance and inadequate decongestion as well as poor prognosis. WRF has been attributed to a reflex renal vasoconstriction elicited by intravascular volume depletion during brisk diuresis. The investigators hypothesize that CHF patients with hepatic dysfunction are more prone to WRF due to poor albumin production. This sub-group of CHF patients may benefit more (increased diuretic efficacy and protected against worsening renal function) by the use of IV loop diuretics in combination with an intravascular volume expander such as IV Human Albumin.

DETAILED DESCRIPTION:
Acute decompensation of chronic heart failure (CHF) warranting hospital admission, defined as diagnosed on the basis of the presence of at least one symptom (dyspnea, orthopnea, paroxysmal nocturnal dyspnea, weight gain, worsening functional class or edema) and one sign (rales, peripheral edema, ascites, increased jugular vein pressure, hepatomegaly, third heart sound gallop or pulmonary vascular congestion on chest radiography) of heart failure plus laboratory or imaging evidence of hepatic dysfunction at randomization

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 yrs
2. acute decompensation of CHF
3. evidence of hepatic dysfunction by laboratory biochemical measurements or imaging (liver ultrasonography)
4. history of CHF with previous use of an oral loop diuretic
5. anticipated need for IV diuretic therapy for at least 72 hours

There is no pre-specified inclusion criterion with respect to ejection fraction

Exclusion Criteria:

1. hemodynamic collapse (at least one of the following: systolic blood pressure (BP) < 90 mmHg, or BP drop by >= 40 mmHg for >= 15 min, with end-organ hypoperfusion; need for inotropes (except of digoxin); need for cardiopulmonary resuscitation).
2. hepatic dysfunction of other than cardiac etiology
3. severe anemia (Hb<8 g/dL)
4. uncontrolled hypertension or hypertensive emergency/urgency
5. pulmonary edema or pulmonary congestion necessitating use of IV vasodilators
6. serum creatinine > 3 mg/dL or glomerular filtration rate (GFR) < 30 ml/min

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of symptoms | From baseline to 72 hours.
  Patient's global assessment of symptoms, measured with the use of a visual-analogue scale (VAS) and quantified as the area under the curve (AUC) of serial assessments.
Change in the serum creatinine level | From baseline to 72 hours.
  Change in the serum creatinine level

SECONDARY OUTCOMES:
Patient-reported dyspnea | From baseline to 72 hours.
  Patient-reported dyspnea (as assessed with the use of a VAS and quantified as the AUC of serial assessments)
Changes in body weight | From baseline to 72 hours.
  Changes in body weight
Length of stay | From baseline to discharge.
  Length of stay
The composite of death, rehospitalization, escalation in treatment or an emergency room visit within 180 days. | From baseline to 180 days from discharge.
  The composite of death, rehospitalization, escalation in treatment or an emergency room visit within 180 days.
Net fluid loss | From baseline to 72 hours
  Net fluid loss

CONTACTS AND LOCATIONS:
Overall Officials: MARIOS VASILEIOS KOUTROULOS, Principal Investigator — University Hospital of Alexandroupolis
Locations (1):
- DUThrace Cardiology Department, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: No